CLINICAL TRIAL: NCT01951937
Title: Fish Intervention and Learning Abilities in German Youths
Brief Title: Fish Intervention and Learning Abilities
Acronym: FINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: National Institute of Nutrition and Seafood Research, Norway (Other Government)
Responsible Party: Principal Investigator, Prof. Berthold Koletzko, Dr med Dr med habil (MD PhD), Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FINS-547
Record Dates: First submitted 2013-09-20; First posted 2013-09-27 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Cognitive Enhancement
Keywords: Cognitive Test; Omega-3 Fatty acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish Meals (Active Comparator): 3 Fish meals per week for 4 months
  Interventions: Dietary Supplement: Fish Meals
- Placebo (Placebo Comparator): Habitual diet
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fish Meals — Meals containing salmon
  Arms: Fish Meals
Dietary Supplement: Placebo — No fish meals
  Arms: Placebo

SUMMARY:
In the FINS study we test - in a randomized non blinded intervention study- the hypothesis that increased intake of salmon will improve cognitive performance of children aged 4 years to 6 years in the Munich area (Germany), who habitually consume little fish.

DETAILED DESCRIPTION:
Long chain polyunsaturated fatty acids (LC-PUFA) of the n-3 series, eicosapentaenoic acid (EPA) and most prominently docosahexaenoic acid (DHA), are considered important for neural development during pre- and postnatal development.

ELIGIBILITY:
Inclusion Criteria:

* 4-6 years

Exclusion Criteria:

* severe illness
* child dislikes fish

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Performance | Change from baseline at 4 months later

SECONDARY OUTCOMES:
Change of cheek cell glycerophospholipids docosahexaenoic and eicosapentaenoic percentage | Change from baseline at 4 months later
Change of red blood cell fatty acids (omega-3 index),plasma phospholipid species and plasma vitamin D3 | Change from baseline at 4 months later
Change of iodine levels in urine | Change from baseline at 4 months later

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Dr med habil, Study Director — Head, Div. Metabolic and Nutritional Medicine Dr. von Hauner Children's Hospital Univ. of Munich Medical Centre - Klinikum d. Univ. München Lindwurmstr. 4, D-80337 Muenchen, Germany
Locations (1):
- Div. Metabolic and Nutritional Medicine Dr. von Hauner Children's Hospital Univ. of Munich Medical Centre, Munich, Bavaria, Germany

REFERENCES:
- [Result] Demmelmair H, Oyen J, Pickert T, Rauh-Pfeiffer A, Stormark KM, Graff IE, Lie O, Kjellevold M, Koletzko B. The effect of Atlantic salmon consumption on the cognitive performance of preschool children - A randomized controlled trial. Clin Nutr. 2019 Dec;38(6):2558-2568. doi: 10.1016/j.clnu.2018.11.031. Epub 2018 Dec 22. PMID 30598384